CLINICAL TRIAL: NCT04449211
Title: The Effectiveness in the Treatment of Long Bone Defect in Adults Using 3D-printed Titanium Alloy Implant
Brief Title: The Effectiveness in the Treatment of Long Bone Defect Using 3D-printed Implant
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cho Ray Hospital (Other)
Collaborators: Commonwealth Scientific and Industrial Research Organisation, Australia (Other Government); 3 Dimensional Tech Vision Limited Company (Unknown)
Responsible Party: Principal Investigator, Hung Do Phuoc, MD, PhD, Associate Professor, Cho Ray Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChoRayH
Record Dates: First submitted 2020-06-22; First posted 2020-06-26 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Bone Loss; Defect Limb
Keywords: bone defect; 3D-printed Titanium alloy implant; Electron Beam Melting; customised implant; patient-specific implant
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Intervention Model Description: Prospective participants with health insurance admitted to the Orthopaedic and Traumatology Department of Cho Ray hospital who get the diagnosis of bone defect greater than 5cm due to trauma or tumour resection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with massive bone defect (Experimental): Adult participants with health insurance regardless of sex having bone defect greater than 5cm due to trauma or tumour resection agree to participate the research.
  The customised 3D-Printed implant is manufactured and undergoes post-processing treatment before being ready for implantation surgery.
  Interventions: Device: Implantation

INTERVENTIONS:
Device: Implantation — Reconstructing the long bone defect with 3D-printed customised Titanium alloy implant
  Other Names: Bone defect implant

SUMMARY:
To evaluate the effectiveness of 3D-printed titanium alloy implants in the treatment of long bone defect in adults

DETAILED DESCRIPTION:
The participant with long bone defect or bone tumor of the extremity is referred to the Radiology Department to have a full CT-scan of both limbs to facilitate the later reconstruction. With the contralateral limb CT-scan data, the implant is designed with appropriate geometry and structures through online meetings with the scientists of CSIRO, Australia. Through this discussion, the supporting guides for the precise osteotomy will also be designed and would be 3D-printed later by 3 Dimensional Tech Vision Limited Company (Vietnam) with Poly Lactic Acid material. The 3D-printed metal parts will be manufactured using Titanium - 6 Aluminum - 4 Vanadium ELI (Extra Low Interstitial) material with Electron Beam Melting technology in CSIRO (Australia). Subsequently, the 3D-printed part will undergo mechanical tests using the Instron 5500R system (Australia) to validate its required mechanical properties. If this metal part cannot fulfill the mechanical requirements, the problematic geometry will be revised and re-designed. Another prototype will be 3D-printed with the same protocol and be tested until it qualified for the mechanical requirement. When the 3D-printed model passes the mechanical test, another 3D-printed metal part with a similar design will be manufactured before transferring to 3-Dimensional Tech Vision Limited Company (Vietnam) for post-processing, surface finishing, sterilising, packaging, labeling. Eventually, the implant will be sent to Cho Ray hospital. The amount of intraoperative blood loss and operative time will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants with health insurance regardless of sex having bone defect greater than 5cm due to trauma or tumour resection agree to participate the research

Exclusion Criteria:

* Participants with contraindication to surgery
* Participants do not agree to undergo surgery
* Participants with local infection or soft tissue defect

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-10-06 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Functional outcome of the upper limb | 1 to 12 months
  For the participant with bone defect of the upper limb, the Disabilities of the Arm, Shoulder, and Hand (DASH) score will be used to evaluate for the limb functional outcome. The scale is ranging from 0 (no disability) to 100 (most severe disability).
Functional outcome of the lower limb | 1 to 12 months
  For the participant with bone defect of the lower limb, the Karlstrom & Olerud score will be used to evaluate for the limb functional outcome. The scale is graded as: bad, fair, good, excellent functional outcome.
Radiological imaging | Post-operative day 1 to 12 months
  the bone healing process is evaluated by the change in dual energy CT-scan result

SECONDARY OUTCOMES:
Complications | through study completion, an average of 1 year.
  Rate of complications

CONTACTS AND LOCATIONS:
Locations (1):
- Cho Ray hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No
Limited data are available only to research providing high quality (of sufficient details as to be useful for research purposes) and accessible (able to be acquired and used) data for research. Those data also include the deidentified data such as X-Ray, CT-scan, MRI, etc. and do not include any identified information

REFERENCES:
- [Background] Nauth A, McKee MD, Einhorn TA, Watson JT, Li R, Schemitsch EH. Managing bone defects. J Orthop Trauma. 2011 Aug;25(8):462-6. doi: 10.1097/BOT.0b013e318224caf0. PMID 21738065
- [Background] Keating JF, Simpson AH, Robinson CM. The management of fractures with bone loss. J Bone Joint Surg Br. 2005 Feb;87(2):142-50. doi: 10.1302/0301-620x.87b2.15874. No abstract available. PMID 15736731
- [Background] Kironde E, Sekimpi P, Kajja I, Mubiri P. Prevalence and patterns of traumatic bone loss following open long bone fractures at Mulago Hospital. OTA Int. 2019 Mar 12;2(1):e015. doi: 10.1097/OI9.0000000000000015. eCollection 2019 Mar. PMID 33937651
- [Background] Le LC, Blum RW. Road traffic injury among young people in Vietnam: evidence from two rounds of national adolescent health surveys, 2004-2009. Glob Health Action. 2013 Jan 17;6:1-9. doi: 10.3402/gha.v6i0.18757. PMID 23336620
- [Background] Ivers RQ, Nguyen HT, La QN. Status of road safety and injury burden: Vietnam. J Orthop Trauma. 2014;28 Suppl 1:S50-1. doi: 10.1097/BOT.0000000000000098. No abstract available. PMID 24858002
- [Background] Masquelet AC, Begue T. The concept of induced membrane for reconstruction of long bone defects. Orthop Clin North Am. 2010 Jan;41(1):27-37; table of contents. doi: 10.1016/j.ocl.2009.07.011. PMID 19931050
- [Background] Iacobellis C, Berizzi A, Aldegheri R. Bone transport using the Ilizarov method: a review of complications in 100 consecutive cases. Strategies Trauma Limb Reconstr. 2010 Apr;5(1):17-22. doi: 10.1007/s11751-010-0085-9. Epub 2010 Mar 9. PMID 20360874
- [Background] Belthur MV, Conway JD, Jindal G, Ranade A, Herzenberg JE. Bone graft harvest using a new intramedullary system. Clin Orthop Relat Res. 2008 Dec;466(12):2973-80. doi: 10.1007/s11999-008-0538-3. Epub 2008 Oct 8. PMID 18841433
- [Background] Cricchio G, Lundgren S. Donor site morbidity in two different approaches to anterior iliac crest bone harvesting. Clin Implant Dent Relat Res. 2003;5(3):161-9. doi: 10.1111/j.1708-8208.2003.tb00198.x. PMID 14575632
- [Background] Robertson PA, Wray AC. Natural history of posterior iliac crest bone graft donation for spinal surgery: a prospective analysis of morbidity. Spine (Phila Pa 1976). 2001 Jul 1;26(13):1473-6. doi: 10.1097/00007632-200107010-00018. PMID 11458153
- [Background] Campana V, Milano G, Pagano E, Barba M, Cicione C, Salonna G, Lattanzi W, Logroscino G. Bone substitutes in orthopaedic surgery: from basic science to clinical practice. J Mater Sci Mater Med. 2014 Oct;25(10):2445-61. doi: 10.1007/s10856-014-5240-2. Epub 2014 May 28. PMID 24865980
- [Background] Roberts TT, Rosenbaum AJ. Bone grafts, bone substitutes and orthobiologics: the bridge between basic science and clinical advancements in fracture healing. Organogenesis. 2012 Oct-Dec;8(4):114-24. doi: 10.4161/org.23306. Epub 2012 Oct 1. PMID 23247591
- [Background] de Alencar PG, Vieira IF. BONE BANKS. Rev Bras Ortop. 2015 Nov 16;45(6):524-8. doi: 10.1016/S2255-4971(15)30297-4. eCollection 2010 Nov-Dec. PMID 27026958
- [Background] Mauffrey C, Barlow BT, Smith W. Management of segmental bone defects. J Am Acad Orthop Surg. 2015 Mar;23(3):143-53. doi: 10.5435/JAAOS-D-14-00018. PMID 25716002
- [Background] Matsuno H, Yokoyama A, Watari F, Uo M, Kawasaki T. Biocompatibility and osteogenesis of refractory metal implants, titanium, hafnium, niobium, tantalum and rhenium. Biomaterials. 2001 Jun;22(11):1253-62. doi: 10.1016/s0142-9612(00)00275-1. PMID 11336297
- [Background] Rotta, G., T. Seramak, and K. Zasińska, Estimation of Young's Modulus of the Porous Titanium Alloy with the Use of Fem Package. Advances in Materials Science, 2015. 15(4): p. 29 - 37
- [Background] Elias, C.N., et al., Biomedical applications of titanium and its alloys. JOM, 2008. 60(3): p. 46-49
- [Background] Heinl P, Muller L, Korner C, Singer RF, Muller FA. Cellular Ti-6Al-4V structures with interconnected macro porosity for bone implants fabricated by selective electron beam melting. Acta Biomater. 2008 Sep;4(5):1536-44. doi: 10.1016/j.actbio.2008.03.013. Epub 2008 Apr 10. PMID 18467197
- [Background] Rho JY, Ashman RB, Turner CH. Young's modulus of trabecular and cortical bone material: ultrasonic and microtensile measurements. J Biomech. 1993 Feb;26(2):111-9. doi: 10.1016/0021-9290(93)90042-d. PMID 8429054
- [Background] Niinomi, M., Mechanical properties of biomedical titanium alloys. Materials Science and Engineering: A, 1998. 243(1): p. 231-236
- [Background] Head WC, Bauk DJ, Emerson RH Jr. Titanium as the material of choice for cementless femoral components in total hip arthroplasty. Clin Orthop Relat Res. 1995 Feb;(311):85-90. PMID 7634595
- [Background] Shi L, Shi L, Wang L, Duan Y, Lei W, Wang Z, Li J, Fan X, Li X, Li S, Guo Z. The improved biological performance of a novel low elastic modulus implant. PLoS One. 2013;8(2):e55015. doi: 10.1371/journal.pone.0055015. Epub 2013 Feb 21. PMID 23437048
- [Background] Stoppie N, Van Oosterwyck H, Jansen J, Wolke J, Wevers M, Naert I. The influence of Young's modulus of loaded implants on bone remodeling: an experimental and numerical study in the goat knee. J Biomed Mater Res A. 2009 Sep 1;90(3):792-803. doi: 10.1002/jbm.a.32145. PMID 18615463
- [Background] Sumner DR, Turner TM, Igloria R, Urban RM, Galante JO. Functional adaptation and ingrowth of bone vary as a function of hip implant stiffness. J Biomech. 1998 Oct;31(10):909-17. doi: 10.1016/s0021-9290(98)00096-7. PMID 9840756
- [Background] Ryan G, Pandit A, Apatsidis DP. Fabrication methods of porous metals for use in orthopaedic applications. Biomaterials. 2006 May;27(13):2651-70. doi: 10.1016/j.biomaterials.2005.12.002. Epub 2006 Jan 19. PMID 16423390
- [Background] Taniguchi N, Fujibayashi S, Takemoto M, Sasaki K, Otsuki B, Nakamura T, Matsushita T, Kokubo T, Matsuda S. Effect of pore size on bone ingrowth into porous titanium implants fabricated by additive manufacturing: An in vivo experiment. Mater Sci Eng C Mater Biol Appl. 2016 Feb;59:690-701. doi: 10.1016/j.msec.2015.10.069. Epub 2015 Oct 28. PMID 26652423
- [Background] Sallica-Leva E, Jardini AL, Fogagnolo JB. Microstructure and mechanical behavior of porous Ti-6Al-4V parts obtained by selective laser melting. J Mech Behav Biomed Mater. 2013 Oct;26:98-108. doi: 10.1016/j.jmbbm.2013.05.011. Epub 2013 May 29. PMID 23773976
- [Background] Dallago M, Fontanari V, Torresani E, Leoni M, Pederzolli C, Potrich C, Benedetti M. Fatigue and biological properties of Ti-6Al-4V ELI cellular structures with variously arranged cubic cells made by selective laser melting. J Mech Behav Biomed Mater. 2018 Feb;78:381-394. doi: 10.1016/j.jmbbm.2017.11.044. Epub 2017 Dec 6. PMID 29220822
- [Background] Vasconcellos LM, Leite DO, Oliveira FN, Carvalho YR, Cairo CA. Evaluation of bone ingrowth into porous titanium implant: histomorphometric analysis in rabbits. Braz Oral Res. 2010 Oct-Dec;24(4):399-405. doi: 10.1590/s1806-83242010000400005. PMID 21180959
- [Background] Chang B, Song W, Han T, Yan J, Li F, Zhao L, Kou H, Zhang Y. Influence of pore size of porous titanium fabricated by vacuum diffusion bonding of titanium meshes on cell penetration and bone ingrowth. Acta Biomater. 2016 Mar;33:311-21. doi: 10.1016/j.actbio.2016.01.022. Epub 2016 Jan 21. PMID 26802441
- [Background] Rybicki, F.J., 3D Printing in Medicine: A Practical Guide for Medical Professionals. 2017: Springer. 1 - 22
- [Background] Zadpoor, A.A., Mechanical meta-materials. Materials Horizons, 2016. 3(5): p. 371-381
- [Background] Imanishi J, Choong PF. Three-dimensional printed calcaneal prosthesis following total calcanectomy. Int J Surg Case Rep. 2015;10:83-7. doi: 10.1016/j.ijscr.2015.02.037. Epub 2015 Mar 10. PMID 25827294
- [Background] Aranda JL, Jimenez MF, Rodriguez M, Varela G. Tridimensional titanium-printed custom-made prosthesis for sternocostal reconstruction. Eur J Cardiothorac Surg. 2015 Oct;48(4):e92-4. doi: 10.1093/ejcts/ezv265. Epub 2015 Aug 4. PMID 26242897
- [Background] Kim D, Lim JY, Shim KW, Han JW, Yi S, Yoon DH, Kim KN, Ha Y, Ji GY, Shin DA. Sacral Reconstruction with a 3D-Printed Implant after Hemisacrectomy in a Patient with Sacral Osteosarcoma: 1-Year Follow-Up Result. Yonsei Med J. 2017 Mar;58(2):453-457. doi: 10.3349/ymj.2017.58.2.453. PMID 28120579
- [Background] Wen X, Gao S, Feng J, Li S, Gao R, Zhang G. Chest-wall reconstruction with a customized titanium-alloy prosthesis fabricated by 3D printing and rapid prototyping. J Cardiothorac Surg. 2018 Jan 8;13(1):4. doi: 10.1186/s13019-017-0692-3. PMID 29310677
- [Background] Lu Y, Chen G, Long Z, Li M, Ji C, Wang F, Li H, Lu J, Wang Z, Li J. Novel 3D-printed prosthetic composite for reconstruction of massive bone defects in lower extremities after malignant tumor resection. J Bone Oncol. 2019 Jan 25;16:100220. doi: 10.1016/j.jbo.2019.100220. eCollection 2019 Jun. PMID 31044134
- [Background] Marco, F.A.d., A.Z. Rozim, and S.R. Piedade, Estabilidade articular do joelho no quadro do
- [Background] Luo W, Huang L, Liu H, Qu W, Zhao X, Wang C, Li C, Yu T, Han Q, Wang J, Qin Y. Customized Knee Prosthesis in Treatment of Giant Cell Tumors of the Proximal Tibia: Application of 3-Dimensional Printing Technology in Surgical Design. Med Sci Monit. 2017 Apr 7;23:1691-1700. doi: 10.12659/msm.901436. PMID 28388595